CLINICAL TRIAL: NCT04922606
Title: Great Saphenous Vein Anatomy at the Proximal Medial Thigh as a Potential Site for Rescue Venous Access
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tobias Kummer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-002859
Record Dates: First submitted 2021-05-07; First posted 2021-06-10 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Anatomy of the GSV for Rescue Peripheral IV Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- US of GSV (Other): Ultrasound of the Great Saphenous Vein
  Interventions: Diagnostic Test: US ot the GSV

INTERVENTIONS:
Diagnostic Test: US ot the GSV — Ultrasound of the Great Saphenous Vein

SUMMARY:
The purpose of this study is to assess the anatomy of the great saphenous vein at the level of the medial thigh in the general population in an effort to categorize this as a reliable target vessel for rescue peripheral IV access.

ELIGIBILITY:
Inclusion Criteria:

- Pediatric and adult Emergency Department patients and employees of all ages from all areas of the emergency department or additional training sites staffed by emergency medicine residents.

Exclusion Criteria:

* Critically ill patients as determined by the Emergency Medicine consultant of record for the patient.
* Legs not accessible due to dressing, wounds, or other factors.
* Overlying cellulitis/soft tissue infection or injury.
* Patients that are prison inmates and patients/patient's surrogates who are unable to give verbal consent/assent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2045-05 (Estimated); Study Completion 2045-05 (Estimated)

PRIMARY OUTCOMES:
Successful visualization of GSV | 12 months
  Number of times the great saphenous vein is identified at the level of the medial distal thigh in the general population using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kummer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No